CLINICAL TRIAL: NCT05113030
Title: Impact of Polycystic Ovary Syndrome on Periodontal Status of Women of Adolescent and Adult Age Groups: A Cross Sectional Study
Brief Title: Impact of PCOS on Periodontal Status of Adolescent and Adult Age Group Women
Status: Completed | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: swati PCOS perio
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome; Gingival Inflammation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group(1st): PERIODONTAL STATUS OF FEMALE PATIENTS WITH PCOS (NEWLY DIAGNOSED) OF ADOLESCENT AGE GROUP WILL BE ASSESSED
  Interventions: Other: PERIODONTAL STATUS OF FEMALE PATIENTS WITH PCOS (NEWLY DIAGNOSED) OF ADOLESCENT AGE GROUP WILL BE ASSESSED
- Test group(2nd): PERIODONTAL STATUS OF FEMALE PATIENTS WITH PCOS (NEWLY DIAGNOSED) OF ADULT AGE GROUP WILL BE ASSESSED
  Interventions: Other: PERIODONTAL STATUS OF FEMALE PATIENTS WITH PCOS (NEWLY DIAGNOSED) OF ADULT AGE GROUP WILL BE ASSESSED

INTERVENTIONS:
Other: PERIODONTAL STATUS OF FEMALE PATIENTS WITH PCOS (NEWLY DIAGNOSED) OF ADOLESCENT AGE GROUP WILL BE ASSESSED — Test group(1st) enrollment criteria in PCOS group will be females of adolescent age newly diagnosed with PCOS, with >16 natural teeth. The diagnosis of PCOS will be according to Rotterdam criteria, and periodontal parameters will be recorded to evaluate periodontal status
  Groups: Test group(1st)
Other: PERIODONTAL STATUS OF FEMALE PATIENTS WITH PCOS (NEWLY DIAGNOSED) OF ADULT AGE GROUP WILL BE ASSESSED — Test group(2 nd) enrollment criteria in PCOS group will be females of adult age newly diagnosed with PCOS, with >16 natural teeth. The diagnosis of PCOS will be according to Rotterdam criteria, and periodontal parameters will be recorded to evaluate periodontal status
  Groups: Test group(2nd)

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy in women, primarily affecting the reproductive system, with substantial collateral negative health effects on metabolic, psychological, and cardiovascular functions. Patients with this syndrome are at higher risk of developing insulin resistance (IR), obesity, dyslipidemia, cardiovascular disease (CVD), and endometrial carcinoma.IR and hyperinsulinemia are responsible for the low-grade chronic systemic inflammation.

Periodontitis, an immuno-inflammatory disease, is a result of interaction between bacterial attack and host inflammatory response, causing inflammation of supporting tissues of the teeth leading to tissue destruction and tooth loss. Chronic low-grade inflammation is emerging as a plausible etiologic mechanism linking periodontal disease and many systemic diseases. Previous cross-sectional studies described a possible relationship between PCOS and periodontitis and the impact of PCOS on gingival inflammation and vice-versa in terms of increased inflammatory markers (hsCRP, IL-6, IL-17 and TNF-α). In PCOS females, there is an alteration of various hormone levels in the body. Female sex steroid hormones play a key role in periodontal disease progression and periodontal and implant wound healing. Human gingiva has the capacity to metabolize hormones such as estrogen and progesterone. Moreover, gingival tissue exhibits receptors for such hormones and it is considered as a target organ for their direct action. These hormones might act on gingival cells by changing the effectiveness of the epithelial barrier to bacterial injury or by affecting the collagen maintenance and repair.

To avoid periodontal implications as these hormonal changes can worsen the vulnerability to plaque-induced periodontal disease. So, present study is going to conduct in females with PCOS and periodontitis at different age groups like adolescent and adult age groups. AIM - Assessment of impact of polycystic ovary syndrome on periodontal status of women of adolescent and adult age groups.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrinopathy in women, primarily affecting the reproductive system, with substantial collateral negative health effects on metabolic, psychologic, and cardiovascular functio ns.

It is a complex disease with characteristics of hyperandrogenism and chronic anovulation (CA) with global prevalence ranging from 2.2% to 26% in Western countries, 2% to 7.5% in China, 6.3% in Sri Lanka,and 9.13% to 36% in India.Patients with this syndrome are at higher risk of developing insulin resistance (IR), obesity, dyslipidemia, cardiovascular disease (CVD), and endometrial carcinoma IR and hyperinsulinemia are responsible for the low-grade chronic systemic inflammation. Periodontitis, an immunoinflammatory disease, is a result of interaction between bacterial attack and host inflammatory response, causing inflammation of supporting tissues of the teeth leading to tissue destruction and tooth loss. It has been suggested as a risk factor for many systemic diseases such as diabetes mellitus, dyslipidemia, obesity, CVDs, rheumatoid arthritis, and respiratory diseases. Chronic low-grade inflammation is emerging as a plausible etiologic mechanism linking periodontal disease and many systemic diseases. Increased concentrations of inflammatory biomarkers (CRP and interleukin -6) have been reported in periodontitis and periodontal treatment helps in decreasing these biomarkers. Timonen P et al. in their cross sectional study demonstrated association of insulin sensitivity with the periodontal infection but they could not draw definite conclusions about the role of reduced insulin sensitivity in the pathogenesis of periodontal infection. Furthermore, Periodontal intervention may improve glycemic control, insulin resistance and serum inflammatory cytokine levels in type II Diabetes patients having chronic periodontitis. Both PCOS and periodontitis has been linked to elevated CRP levels, therefore it is postulated that CRP might be a possible mediator of the association between periodontitis and PCOS As, periodontitis and PCOS are associated with systemic inflammation and insulin resistance, these two disorders may be linked through a common pathophysiologic pathway. Previously conducted cross-sectional studies described a possible relationship between PCOS and periodontitis and the impact of PCOS on gingival inflammation and vice-versa in terms of increased inflammatory markers (hsCRP, IL-6, IL-17 and TNF-α). However, they have not evaluated the effect of periodontal therapy on systemic inflammation and insulin resistance in PCOS women suffering with periodontitis. It was hypothesized that periodontitis and insulin resistance may add to the systemic inflammatory burden and may consequently contribute to progression of PCOS and vice -versa. So, controlling systemic inflammatory burden by scaling and root planing and medical treatment may have an effect in the management of PCOS women ha ving periodontitis. Therefore, the study was attempted to evaluate the effect of non-surgical periodontal therapy along with medical treatment on hsCRP, Homeostatic Model Assessment (HOMA) and periodontal parameters in PCOS women having periodontitis. Available evidence suggests that oxidative stress may be a common link for the association between periodontitis and components of the metabolic syndrome, diabetes, and CVD. Both nitrites and nitrates, which appear in nitric oxide (NO) metabolism, and myeloperoxidase (MPO) are considered to reflect the strength of oxidative stress.

AIM - assessment of impact of polycystic ovary syndrome on periodontal status of women of adolescent and adult age groups. A cross-sectional study PRIMARY OBJECTIVES Comparative evaluation of periodontal parameters like Bleeding on probing(BOP), probing pocket depth(PPD), clinical attachment level(CAL)in both groups. Comparative evaluation of serum hsCRP levels( high sensitivity C reactive proteins) in both the groups. SECONDARY OBJECTIVES Assessment of Plaque index, Gingival index, Gingival phenotype, Gingival recession, Education status, Socio-economic status, Anthropometric parameters. Objectives Outcome Method of measurement of outcome Comparative evaluation of periodontal parameters( BOP, PD, CAL,PI, GI) in both the groups.

The present cross-sectional study will be conducted in the Department of periodontology, Post Graduate Institute of Dental Sciences, Rohtak in collaboration with Department of Obstetrics and Gynaecology Post Graduate Institute of Medical Sciences, Rohtak

1.PLAQUE INDEX(PI)- Plaque index by Silness and Loe 43(1964) will be used for assessment of plaque. For the scoring, a mouth mirror, an explorer and a light source will be used on air dried teeth and gingiva. GINGIVAL INDEX (GI) : Lӧe and Silness-Gingival Index by Loe and Silness (1963) will be used. 3.BLEEDING ON PROBING (BOP):BOP will be recorded as 1 (present) if it occurred within 15 sec of probing and 0 (absent) if no bleeding occurred. It will be calculated in %.

After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100. It will be designed as % sites with bleeding on probing. 4.PROBING POCKET DEPTH (PPD):Probing pocket depth will be measured as the distance from the gingival margin to the base of the clinical pocket. The probing depth measurements will be assessed using a calibrated manual periodontal probe (PCP-UNC 15Hu-Friedy, Chicago, IL, USA).

5. CLINICAL ATTACHMENT LEVEL (CAL): Clinical Attachment Level will be measured as the distance between the base of the clinical pocket and the cemento-enamel junction(CEJ).Measurements will be made at 6 sites of involved tooth- mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual using UNC-15 probe. Measurements will be rounded to the nearest whole millimetre. Distance of base of the pocket from gingival margin, distance of free gingival margin from CEJ. 6. Gingival health (According to AAP,2017 classification) 7. Gingivitis (Dental plaque induced)-According to AAP,2017 classification

8.SURVEILLANCE OF PERIODONTITIS( According to AAP,2017 classification) Radiographs (if needed) for evaluation of staging and grading of periodontitis. (According to AAP, 2017 classification) 9. Gingival phenotype Thin scalloped biotype in which there is a greater association with slender triangular crown, subtle cervical convexity, interproximal contacts close to the incisal edge and a narrow zone of KT, clear thin delicate gingiva, and a relatively thin alveolar bone.

Thick flat biotype showing more square-shaped tooth crowns, pronounced cervical convexity, large interproximal contact located more apically, a broad zone of KT, thick, fibrotic gingiva, and a comparatively thick alveolar bone. Thick scalloped biotype showing a thick fibrotic gingiva, slender teeth, narrow zone of KT, and a pronounced gingival scalloping. 10. Gingival recession It is defined as the apical shift of the gingival margin with respect to the cemento-enamel junction (CEJ); it is associated with attachment loss and with exposure of the root surface to the oral environment

Cairo, 2011:

According to American Academy of Periodontology and European Federation of Periodontology,2017 classification. 11. Analyses of Anthropometric Parameters,Waist circumference (WC) will be measured in centimetres, at the midpoint between the lower margin of the lowest palpable rib and the top of the iliac crest. For waist-to-hip ratio (WHR), hip circumference will be measured around the widest portion of the buttocks. BMI(Kg/m²) will be recorded as weight in kilograms divided by height in meters squared. 12.Blood Sampling- Blood samples for the investigation of serum hsCRP will be collected after overnight fasting. Venous blood from the antecubital vein will be collected after applying a tourniquet in plain tubes without additive. Serum hsCRP levels will be assessed using a kit‡ with high sensitivity methodology in an auto-analyzer§ according to the manufacturer's instructions. The test principle will be particle-enhanced immune-turbidimetric assay, in which human CRP agglutinates with latex particles coated with monoclonal anti-CRP antibodies. The turbidity induced by the formation of immune complexes will be measured at 546 nm.

The lower detection limit for the assay was 0.15 mg/L. Serum Testosterone levels (if required) 13. PCOSQ (Polycystic ovary syndrome questionnaire)- Given by Cronin et al. for psychological status and quality of life. 14. Phenotype of PCOS- According to Rotterdam criteria and AE-PCOS Society criteria.

ELIGIBILITY:
Inclusion Criteria-

* females of adolescent and adult age groups newly diagnosed with PCOS(according to Rotterdam criteria), with >16 natural teeth.
* age range (11-19Year) for adolescent age group
* age range (20-40Year) for adult age group..

Exclusion Criteria:

* Patients with any history of thyroid dysfunction, hyperprolactinemia and androgen-secreting tumors to avoid misdiagnosis of PCOS.
* Patients with chronic inflammatory disease such as nephrotic syndrome, chronic renal failure, significant cardiovascular disease, established type 1 or type 2 diabetes mellitus, or active cancer within the past 5 years will be excluded to control the confounders. With history of substance abuse (Tobacco/Alcohol) History of systemic antibiotics within 3 months Periodontal treatment within 6 months Aggressive periodontitis cases Females on oral contraceptive pills, pregnancy, lactation.

Ages: 11 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: females of adolescent and adult age groups newly diagnosed with PCOS without taking treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing(BOP), | 6 months
  BOP will recorded as 1 (present) if bleeding occur within 15 sec of probing and 0 (absent) if no bleeding occurred. It will be calculated in %
Probing pocket depth(PPD), in both the groups. | 6 months
  The distance from the gingival margin to the base of the clinical pocket.
Serum hsCRP levels( high sensitivity C reactive proteins) | 6 months
  Serum hsCRP levels were assessed using a kit with high sensitivity methodology in an auto-analyzer according to the manufacturer's instructions. The test principle was particle-enhanced immune-turbidimetric assay, in which human CRP agglutinates with latex particles coated with monoclonal anti-CRP antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: SWATI Jaglan, Principal Investigator — Post graduate institute of dental sciences,Rohtak,Haryana
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India